CLINICAL TRIAL: NCT02266771
Title: Impact of V.A.C. Veraflo Therapy in Wounds Requiring Debridement Within an Orthopedic Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBridge Health (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2169
Record Dates: First submitted 2014-09-24; First posted 2014-10-17 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Wounds and Injuries
Keywords: Negative Pressure Wound Therapy, Wound VAC, Instillation
MeSH Terms: conditions — Wounds and Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPWT with Instillation (Active Comparator): Negative Pressure Wound Therapy with Instillation.
  Interventions: Device: NPWT with Instillation
- NPWT without Instillation (Placebo Comparator): Negative Pressure Wound Therapy without Instillation
  Interventions: Device: NPWT

INTERVENTIONS:
Device: NPWT with Instillation — Kinetic Concepts Inc. V.A.C Ulta Negative Pressure Wound Therapy System with V.A.C. VeraFlo Instillation
  Arms: NPWT with Instillation
Device: NPWT — Kinetic Concepts Inc. V.A.C Ulta Negative Pressure Wound Therapy System
  Arms: NPWT without Instillation

SUMMARY:
The objective to this study is to determine the effectiveness of V.A.C.Veraflo negative pressure wound therapy with instillation, when compared to historical controls of V.A.C Therapy without instillation in the management of wounds.

DETAILED DESCRIPTION:
The V.A.C.Ulta™ Negative Pressure Wound Therapy System is a 510(k) -cleared, Class II device (K100657) with the following indication for use: "the V.A.C.Ulta™ Negative Pressure Wound Therapy System is an integrated wound management system that provides Negative Pressure Wound Therapy with an instillation option. Negative Pressure Wound Therapy in the absence of instillation is intended to create an environment that promotes wound healing by secondary or tertiary (delayed primary) intention by preparing the wound bed for closure, reducing edema, promoting granulation tissue formation and perfusion, and by removing exudates and infectious material. The instillation option is indicated for patients who would benefit from vacuum assisted drainage and controlled delivery of topical wound treatment solutions and suspensions over the wound bed. The V.A.C.Ulta™ Negative Pressure Wound Therapy System, with and without instillation, is indicated for patients with chronic, acute, traumatic, sub-acute and dehisced wounds, partial-thickness burns, ulcers (such as diabetic, pressure and venous insufficiency), flaps and grafts". The V.A.C. Ulta™ Therapy Unit is for use with only V.A.C.® Dressings (V.A.C.® GranuFoam™, V.A.C. GranuFoam Silver®, V.A.C. WhiteFoam,® V.A.C. VeraFlo™ Dressing Systems) and disposables. The V.A.C. VeraFlo™ Dressing System is intended for use with V.A.C. VeraFlo™ Therapy as provided by the V.A.C.Ulta™ Therapy Unit. The V.A.C. VeraFlo™ Dressing was cleared under the V.A.C Ulta™ Negative Pressure Wound Therapy System 510(k) (K100657). It is recommended for use with open wounds, including wounds with shallow undermining or tunnel areas where the distal aspect is visible.

Prontosan® Wound Irrigation Solution is a clear, odorless, colorless solution consisting of polyhexamethylene biguanide (PHMB), betaine, sodium hydroxide and purified water. PHMB, also known as Polyhexanide, is a polymer biguanide. PHMB is a cationic preservative which inhibits the growth of microorganisms within the product. Betaine is a zwitterionic (both, negatively and positively charged) surfactant. Prontosan® is a FDA 510(k) cleared device intended for cleaning wounds and for moistening and lubricating absorbent wound dressings for ulcers, burns, post surgical wounds, and abrasions.

The objective to this study is to determine the effectiveness of V.A.C.Veraflo negative pressure wound therapy with Prontosan instillation, when compared to historical controls of V.A.C Therapy without instillation in the management of wounds. We will measure any difference in length of hospital stay, number of days until final surgical procedure, and the number of trips to the or for additional debridement. Patients will be considered infection free when clinical signs of infection are absent and lab values become normal.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent.
* Patients requiring surgical debridement for wounds with exposed hardware and/or bone, traumatic wounds, dehisced wounds, post-surgical wounds, and pressure ulcers/sores requiring debridement.
* Age: 18 years and above.
* Gender: Male or Female.
* No use of Investigational Agents/Devices on study or within 30 days prior to enrollment.
* Subjects who will be locally available for the next 6 months.

Exclusion Criteria:

* Wounds involving prosthetic joints.
* Patients who are unable to adhere to scheduled study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of days between the initial and final surgical procedure. | 6 months

SECONDARY OUTCOMES:
Length of hospital stay | 6 months
Number of days until wound closure | 6 months
Number of operative debridements | 6 months
Recurrence of wound post discharge | 30 days
Wound related re-admission | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Janet D Conway, MD, Principal Investigator — Rubin Institute for Advanced Orthopedics, Sinai Hospital of Baltimore, LifeBridge Health
Locations (1):
- Rubin Institute for Advanced Orthopedics, Sinai Hospital of Baltimore, LifeBridge Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No